CLINICAL TRIAL: NCT07253922
Title: A Prospective Evaluation of Optic Nerve Sheath Diameter Changes Measured by Ultrasonography During Cardiopulmonary Bypass in Patients Undergoing Open Heart Surgery
Brief Title: Evaluation of Optic Nerve Sheath Diameter Changes During Cardiopulmonary Bypass in Open Heart Surgery
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Burak Omur, Assistant Professor of Anesthesiology, Medipol University
Other Study IDs: Medipol-OSKC-2025
Record Dates: First submitted 2025-08-22; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Open Heart Surgery; Cardiopulmonary Bypass; Intracranial Pressure; Optic Nerve Sheath Diameter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: Adult patients (18-85 years) undergoing elective open-heart surgery with cardiopulmonary bypass. Optic nerve sheath diameter (ONSD) will be measured by ultrasonography at predefined time points, along with hemodynamic parameters, NIRS values, and arterial blood gas analyses.
  Interventions: Procedure: Ultrasonography of the Optic Nerve Sheath

INTERVENTIONS:
Procedure: Ultrasonography of the Optic Nerve Sheath — Ultrasonographic measurement of the optic nerve sheath diameter (ONSD) will be performed using a 7.5 MHz linear probe. Measurements will be taken 3 mm behind the globe in both transverse and sagittal planes, three times for each eye, and the average value will be recorded at predefined time points during cardiopulmonary bypass.

SUMMARY:
During cardiopulmonary bypass (CPB) in open-heart surgery, direct measurement of intracranial pressure is not feasible. Evaluation of the optic nerve sheath diameter (ONSD) by ultrasonography is considered a reliable method for predicting increases in intracranial pressure. This study aims to investigate changes in ONSD in patients undergoing open-heart surgery with CPB.

DETAILED DESCRIPTION:
Several mechanisms during CPB-including inflammatory response, hemodilution, reperfusion injury, hypothermia-rewarming imbalances, and microembolism formation-can lead to increased intracranial pressure and cerebral edema. Ultrasonographic measurement of ONSD provides a noninvasive means of monitoring these changes. In this study, ONSD will be measured at different time points, while hemodynamic parameters, NIRS values, and arterial blood gas analyses will be recorded simultaneously. The primary objective is to evaluate changes in ONSD, and the secondary objective is to determine the potential impact of these changes on intracranial pressure.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-85 years
* Scheduled for elective open-heart surgery with cardiopulmonary bypass
* Provided written informed consent

Exclusion Criteria:

* Ocular or neurological complications related to diabetes
* History of previous eye, brain, or thoracic surgery
* Diagnosis of hydrocephalus, glaucoma, intracranial mass, or stroke

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (18-85 years) undergoing elective open-heart surgery with cardiopulmonary bypass at Istanbul Medipol University Hospital, who meet inclusion criteria and provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Change in Optic Nerve Sheath Diameter (ONSD) | From tracheal intubation (baseline) until the end of surgery (approximately 4-6 hours); measurements at six predefined time points (post-intubation, CPB initiation, 15 min, 45 min, 15 min after CPB termination, end of surgery).
  Evaluation of ONSD changes measured by ultrasonography to assess potential alterations in intracranial pressure during cardiopulmonary bypass.

SECONDARY OUTCOMES:
Mean Arterial Pressure (MAP) | From induction of anesthesia until the end of surgery, recorded simultaneously with OSD measurements.
  Measurement of mean arterial pressure.
Central Venous Pressure (CVP) | From induction of anesthesia until the end of surgery, recorded simultaneously with OSD measurements.
  Measurement of central venous pressure.
Arterial Blood pH | From tracheal intubation (baseline) until the end of surgery (approximately 4-6 hours); measurements at six predefined time points (post-intubation, CPB initiation, 15 min, 45 min, 15 min after CPB termination, end of surgery).
  Analysis of arterial blood pH values
Partial Pressure of Arterial Carbon Dioxide (PaCO₂) | From tracheal intubation (baseline) until the end of surgery (approximately 4-6 hours); measurements at six predefined time points (post-intubation, CPB initiation, 15 min, 45 min, 15 min after CPB termination, end of surgery).
  Analysis of partial pressure of arterial carbon dioxide.
Lactate | From tracheal intubation (baseline) until the end of surgery (approximately 4-6 hours); measurements at six predefined time points (post-intubation, CPB initiation, 15 min, 45 min, 15 min after CPB termination, end of surgery).
  Analysis of blood lactate levels.
partial Pressure of Arterial Oxygen (PaO₂) | From tracheal intubation (baseline) until the end of surgery (approximately 4-6 hours); measurements at six predefined time points (post-intubation, CPB initiation, 15 min, 45 min, 15 min after CPB termination, end of surgery).
  Analysis of partial pressure of arterial oxygen.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Omur B, Ciftci B, Karaaslan P. Evaluation of optic nerve sheath diameter in patients undergoing laparoscopic surgery in the Trendelenburg position: a prospective observational study. Ann Saudi Med. 2024 Sep-Oct;44(5):319-328. doi: 10.5144/0256-4947.2024.319. Epub 2024 Oct 3. PMID 39368121
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):e38-360. doi: 10.1161/CIR.0000000000000350. Epub 2015 Dec 16. No abstract available. PMID 26673558
- [Background] Ismail A, Semien G, Sharma S, Collier SA, Miskolczi SY. Cardiopulmonary Bypass. 2024 Aug 12. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482190/ PMID 29489210